CLINICAL TRIAL: NCT04269161
Title: NICU Oxygen Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Sacred Heart Health System (Other)
Responsible Party: Principal Investigator, Roger C Fales, Associate Professor of Mechanical and Aerospace Engineering, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2003117
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Hyperoxia; Hypoxia
MeSH Terms: conditions — Hyperoxia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Crossover Sequence 1 (Experimental): In this arm, an automatic oxygen control device will be used to make adjustments to the blend of oxygen and air supplied to the subject for the first six hours.
  In this arm, a nurse will manually make adjustments to the blend of oxygen and air supplied to the subject for the second six hours. The study continues in an automatic and manual repeating pattern for six days.
  Interventions: Device: Automatic control of inspired oxygen
- Crossover Sequence 2 (Experimental): In this arm, a nurse will manually make adjustments to the blend of oxygen and air supplied to the subject as in the standard of care for the first six hours.
  In this arm, an automatic oxygen control device will be used to make adjustments to the blend of oxygen and air supplied to the subject for the second six hours. The study continues in a manual and automatic repeating pattern for six days.
  Interventions: Device: Automatic control of inspired oxygen

INTERVENTIONS:
Device: Automatic control of inspired oxygen — A device will be used to automatically adjust the blend of oxygen and air with the ability to return to manual control as needed.

SUMMARY:
Prematurely born infants in the hospital neonatal intensive care unit (NICU) will be included in the study. This clinical trial is a randomized crossover study to show that our automated oxygen control device performance is no worse than a NICU nurse in keeping a premature neonate's SPO2 within the prescribed range. Since subjects receive the device (automatic oxygen control) and the standard of care (manual control by a nurse), every subject serves as their own perfectly matched control. Performance measures include the average time it takes for the SpO2 to return to the desired range (primary endpoint) and the total amount of time that the SpO2 is within the desired range (secondary endpoint). The device will be applied to premature infants on respiratory support humidified high flow nasal cannula (HFNC) with oxygen controlled using a blend valve. Two groups include one that begins the study period with the device and one that begins the study period without the device. The two groups are switched between manual and automatic every 6 hours into the trial period and complete a total of 6 days. The target number of subjects is 60. We will analyze the study as a superiority trial if there is strong evidence of superiority.

DETAILED DESCRIPTION:
We intend to enroll between 20-30 subjects at each of two separate institutions (University of Missouri Women's and Children's Hospital and Studer Family Children's Hospital in Pensacola, FL). The subjects will be premature infants <34 weeks post conceptual age (PCA) requiring respiratory support. This randomized clinical trial will utilize a 24 period 2 treatment crossover design to show that the device performs no worse than (non-inferiority trial) an NICU nurse in keeping a premature neonate's SpO2 within the prescribed range while the infant is on respiratory support. Due to the nature of the study, any masking of the intervention is not possible. Upon enrollment, the subjects will be randomized into enrollment in two groups (A and B). The primary endpoint will be the mean time required to re-establish SpO2 within the prescribed range, as measured from the time an out-of-range alarm is triggered. A secondary endpoint will be proportion of time SpO2 is within the prescribed range, using an area-under-the-curve approach (with a discrete state) to account for varying time-on-test. These outcome measures are complementary because the former doesn't account for the number of alarms, while the latter does. This is important because the oxygen control device operates continuously in a proactive manner, rather than only reacting due alarms, so it is doing more than mimicking the nurse -- the second measure allows us to capture that.

Group A will initially have the automatic device interface with HFNC for 6 hours. The device will have the target SpO2 parameters ordered by the treating physician input into the device. A study laptop will interface with the device, cardiopulmonary monitor, and pulse oximeter to record the data for the study. Sensors will be used to record all adjustments to the device/respiratory support equipment (i.e. blend valve and flow valve used in HFNC). These sensors will continuously record the data for later analysis. The device will constantly evaluate data sent to it from the pulse oximeter and bedside monitor recording all of the data and alarms. In response to alarms, displayed data, doctor's orders, etc., nurses will continue to apply manual inputs to make adjustments to flow and provide tactile stimulus to the subject but not adjust FiO2 unless manual mode is selected. Recorded sensor measurements and manual inputs by the nurse will be used to refine the existing models as well as new models of response in HR, RR, and SpO2 to flow adjustments and tactile stimulus.

After the first 6 hours, the device will be switched to manual mode for the subject (nurse makes all adjustments for FiO2), but the laptop and sensor data logging system will continue to record data from the patient and the respiratory support equipment. This will record the information for the nurse intervention/baseline care part of the study, which continue for 6 hours. During the entire process, the bedside nurse will keep a diary of any events/interventions using the time prominently displayed on the monitoring laptop. This "time-stamped" diary system will allow for easier retrieval of and comparison to the data from the device and monitoring laptop. Also, the monitoring laptop will have a record of all the data, including alarms from the pulse oximeter as well as the bedside monitor to allow for easier retrieval of data related to alarm events and interventions. The laptop will also record any interventions made by the device to allow for easier retrieval of data related to device interventions. The treatment will then alternate periods of each treatment for a total of 6 days (24 6-hour periods).

Group B will have the exact opposite order as group A. Group B infants will initially have the laptop interface with all of the monitors and sensor measurements. However, the nurse intervention/baseline care stage of the study will take place for the first 6 hours. Next, group B will have the device interface with their respiratory equipment, and the data will be recorded as described above for the next 6 hours of the study. The the treatment will alternate every 6 hours for a total of 6 days.

This design was chosen because the premature infants should have fewer events as they grow older each day, and it will help take into account this potential bias. Also, the subjects will be randomized to group A or B in sets of 8 (i.e. in each group of 8 envelopes, 4 will be group A and 4 will be group B). During the entire study process the infants will receive normal NICU care and the parameters for the SpO2 range will be set by the physician caring for the infant. There are also built in manual overrides for the device which allow the NICU to make changes while the subject is on the device phase of the study. The device will be able to record these changes and the staff will record their manual interventions in the study diary.

We have planned our sample size using a non-inferiority test for a cross-over design, based on our primary endpoint, t_delta. For a given patient, define t_delta = (mean elapsed time needed for device to re-establish SpO2 after alarm) - (mean elapsed time needed for nurse to re-establish SpO2 after alarm). The margin of non- inferiority will be chosen as t_delta > -10 sec, so that a device which is no worse than 10 sec, on average, than a nurse will be considered non-inferior. Assuming the standard deviation of t_delta =12 and the true mean difference is zero under the alternate hypothesis, a sample size of 48 achieves 88% with alpha=0.05. If there is 16% patient drop-out before crossover, so that the final n=40, the power drops to 82%. In all analysis, a (paired) t-test will be used. Our secondary endpoint is secondary endpoint is the proportion of time SpO2 is within the prescribed range, using an area-under-the-curve approach (with a discrete state) to account for varying time-on-test. Our secondary endpoint will be analyzed in a similar manner.

We will plan for one interim analysis to determine if the trial should be stopped early due to futility (strong evidence of inferiority, where a confidence interval for t_delta lies entirely to the left of -10 and doesn't intersect -10) or for efficacy (strong evidence of superiority with margin > +20 sec). This will be carried out when n=32 (16 subjects per site) is attained and stopping decisions will be based on O'Brien-Fleming stopping principles. The interim analysis will be carried out by an independent statistician on the University of Missouri's Data Safety and Monitoring Committee, which is also available to monitor the study for adverse events if requested by the IRB. In the event that the patient drop-out is greater than 16% before crossover, then a more complicated estimation procedure will be employed using mixed effects models; otherwise, complete cases will be used.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU
* Less than 31 weeks estimated gestational age or less than 1500 grams at birth
* Currently on high flow nasal cannula or bubble CPAP
* Require at least 2 adjustments to the FiO2 per shift and/or have at least 2 desaturation events per shift

Exclusion Criteria:

* Infants admitted to the NICU with congenital heart disease.
* Infants who are set on a minimum FiO2 set point by their healthcare provider

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Pardalos, MD, Principal Investigator — University of Missouri-Columbia; Ramak R Amjad, MD, Principal Investigator — Studer Family Children's Hospital at Sacred Heart; Roger C Fales, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Studer Family Children's Hospital at Sacred Heart, Pensacola, Florida
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou X, Faqeeh A, Amjad R, Pardalos J, Fales R. Clinical Evaluation of an Automatic Oxygen Control System for Premature Infants Receiving High-Flow Nasal Cannula for Respiratory Support: A Pilot Study. J Med Device. 2022 Sep 1;16(3):031005. doi: 10.1115/1.4054250. Epub 2022 May 10. PMID 35646226

RESULTS

PARTICIPANT FLOW:
Groups:
- Crossover Sequence 1: In this arm, an automatic oxygen control device will be used to make adjustments to the blend of oxygen and air supplied to the subject for the first six hours.
  In this arm, a nurse will manually make adjustments to the blend of oxygen and air supplied to the subject for the second six hours. The study continues in an automatic and manual repeating pattern for six days.
  Automatic control of inspired oxygen: A device will be used to automatically adjust the blend of oxygen and air with the ability to return to manual control as needed.
- Crossover Sequence 2: In this arm, a nurse will manually make adjustments to the blend of oxygen and air supplied to the subject as in the standard of care for the first six hours.
  In this arm, an automatic oxygen control device will be used to make adjustments to the blend of oxygen and air supplied to the subject for the second six hours. The study continues in a manual and automatic repeating pattern for six days.
  Automatic control of inspired oxygen: A device will be used to automatically adjust the blend of oxygen and air with the ability to return to manual control as needed.
Period: Overall Study
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2
Started | 24 | 24
Completed | 19 | 20
Not Completed | 5 | 4
Not completed — Change of modality and no longer eligible | 3 | 3
Not completed — Required procedure outside of NICU | 1 | 0
Not completed — Equipment issue | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data from 39 participants completing six days of the study evaluated for the recruitment period.
Groups:
- Crossover Sequence 1 and 2, Automatic, Manual and Manual, Automatic: This group is comprised of Crossover Sequence 1 and Crossover Sequence 2 with all participants that completed six days in the study.
  The automatic oxygen control device or the nurse made adjustments to the blend of oxygen and air supplied to the participant for alternating blocks of six hours.
  The study continues in an automatic and manual repeating pattern for six days.
Arm/Group | Crossover Sequence 1 and 2, Automatic, Manual and Manual, Automatic
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: days] — Age at start of study in days.
  days | 42.897 (27.649)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age at birth in weeks.
  weeks | 27.428 (2.448)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 30
  More than one race | 2
  Unknown or Not Reported | 0
Crossover Sequence 1 or 2 [Count of Participants; unit: Participants]
  Sequence 1 - Automatic, Manual | 19
  Sequence 2 - Manual, Automatic | 20
Modality [Count of Participants; unit: Participants]
  High-Flow Nasal Cannula (HFNC) | 22
  Bubble CPAP (BCPAP) | 17
Weight at start of study [Mean (Standard Deviation); unit: grams] | 1702.205 (531.817)
Bed type [Count of Participants; unit: Participants]
  Isolette | 32
  Open Crib | 7

OUTCOME MEASURES:

1. Primary Outcome: Elapsed Time to Respond to SpO2 Alarm
Description: Mean in elapsed time needed to re- establish SpO2 within the desired range after an alarm. The alarms and alarm times are recorded directly from the bedside monitor and the responses are measured directly in terms of the blend valve position and SpO2 response measured by the pulse oximeter.
Time Frame: Twenty-four study periods consisting of 6-hour manual study periods and 6-hour automatic study periods over six days for each of the subjects in the analysis.
Population: All participants that completed six days of the crossover study period were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Manual Mode (Nurse): Nurse adjusts the blend of oxygen and air manually for six hour periods (no automatic oxygen control by the device).
- Automatic Mode (Device): An investigational device used to automatically adjust the blend of oxygen and air for six-hour periods with the ability to return to manual control as needed.
Arm/Group | Manual Mode (Nurse) | Automatic Mode (Device)
Number analyzed (Participants) | 39 | 39
seconds | 51.408 (66.168) | 41.523 (30.771)
Statistical Analysis 1: Comparison: Manual Mode (Nurse) vs Automatic Mode (Device); A sample requirement of 48 patients was determined based on a pilot study to provide 88% power, and 0.05 significance (two sided) to show the mean difference is less than 10 seconds based on a 2x2 crossover design. Considering patient drop-out, a sample size of n=40 drops power to 82%; Test type: Non-Inferiority — The margin of non-inferiority is 10 seconds such that the device is no worse than 10 seconds on average than manual mode. Our study is a 2-treatment, 24-period crossover design that accounts for first-order carryover effects, indicating a slightly higher power than a 2x2. Each subject acted as their own control. The study was defined as intention to treat, such that manual adjustments during the automated arm would be included in that arm; p = 0.003, t-test, 2 sided — The p-value is significant at 0.01; Mean Difference (Net) = -9.885, 95% CI 2-sided [-16.51 to -3.27] — The difference is time to re-establish in automatic mode minus time to re-establish in manual mode. (a negative number favors automatic mode)

2. Secondary Outcome: Proportion of Time SpO2 is Within the Prescribed Range in a Six-hour Time Block
Description: For each 6-hour time block, we calculate the proportion of time the patient stays within the prescribed SpO2 range. The proportion of time that the SpO2 is within the prescribed range is computed using an area-under-the-curve approach for data taken during automatic control by the experimental device and manual control by the nurse.
Time Frame: Twelve 6-hour manual study periods and 6-hour automatic study periods over six days for each of the subjects in the analysis.
Population: All participants who completed six days in the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: proportion of time
Groups:
- Manual Mode (Nurse): Nurse adjusts the blend of oxygen and air manually for six-hour periods (no automatic oxygen control by the device).
- Automatic Mode (Device): A device used to automatically adjust the blend of oxygen and air for six-hour periods with the ability to return to manual control as needed.
Arm/Group | Manual Mode (Nurse) | Automatic Mode (Device)
Number analyzed (Participants) | 39 | 39
proportion of time | 0.676 (0.214) | 0.695 (0.224)
Statistical Analysis 1: Comparison: Manual Mode (Nurse) vs Automatic Mode (Device); The difference in the proportion of time in the target saturation is calculated between the automatic and manual models. For each 6-hour time block, we calculate the proportion of time the patient stays within the prescribed SpO2 range; Test type: Other — The difference is defined as the difference of proportion of time in the target range of SpO2 in modes, automatic minus manual. Our study is a 2-treatment, 24-period crossover design that accounts for first-order carryover effects, indicating a slightly higher power than a 2x2. Each subject acted as their own control. The study was defined as intention to treat, such that manual adjustments during the automated arm would be included in that arm; p = .02, t-test, 2 sided — The threshold for statistical significance is p=.05; Two-sample t test with equal variances. Linear mixed model patient random effects, adjusted for site, sex, race, weight, gestational age, bed type; Mean Difference (Net) = .018, 95% CI 2-sided [0.003 to .034] — Treatment difference = automatic - manual. A positive number favors automatic

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the, up to, six-day experimental crossover period for each participant in the study.
Arm/Group | Manual Mode (Nurse) | Automatic Mode (Device)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2023-05-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT04269161/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT04269161/SAP_001.pdf
  • Informed Consent Form: Consent 1, Missouri (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04269161/ICF_002.pdf
  • Informed Consent Form: Consent 2, Florida (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04269161/ICF_003.pdf